CLINICAL TRIAL: NCT02061995
Title: Treatment of Severe Osteoporosis by Intravenous Infusion of Pre-osteoblastic Cells - An Open Pilot Study
Brief Title: Phase 2a Study on Intravenous Infusion of Autologous Osteoblastic Cells in Severe Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PREOB-OP1
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2014-02

CONDITIONS: Severe Osteoporosis
Keywords: Bone Diseases; Metabolic Bone Diseases; Osteoporosis; Bone Fractures; Osteoporotic Fractures; Musculoskeletal Diseases
MeSH Terms: conditions — Osteoporosis; Bone Diseases; Bone Diseases, Metabolic; Fractures, Bone; Osteoporotic Fractures; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PREOB® Intravenous Infusion (Experimental)
  Interventions: Drug: PREOB® Intravenous Infusion

INTERVENTIONS:
Drug: PREOB® Intravenous Infusion — Each patient will undergo a single intravenous administration of PREOB®.

SUMMARY:
Osteoporosis is a systemic skeletal disease characterized by low bone mass and microarchitectural deterioration of bone tissue, with a subsequent increase in bone fragility and susceptibility to fracture.

Osteoporosis is one of the most common and debilitating chronic diseases, and a global health concern with a high prevalence not only in Western countries, but also in Asia and Latin America. Most efficacious anti-osteoporotic treatments either inhibit bone resorption like bisphosphonates or denosumab or increase bone formation like teripartide an anabolic agent. Anti-osteoporotic drugs have demonstrated safety and efficacy with an increase in bone mass and a decrease of fracture risk (at the hip) by 30 to 50% after 3 years of treatment (Black et al., 1996; Neer et al., 2001; Meunier et al., 2004). Despite the availability of pharmacological treatments, osteoporosis remains a significant health problem for patients who do not respond to the available treatments or fail to comply with their regimens.

The present phase 2a study aims to demonstrate the safety and efficacy of PREOB®, a proprietary population of autologous osteoblastic cells, in the treatment of osteoporotic patients who do not respond to pharmacological treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe osteoporosis
* Non-response to anti-osteoporotic treatment for over 2 years
* Normal hematology function
* Ability to provide a written, dated, and signed informed consent prior to any study related procedure, and to understand and comply with study requirements

Exclusion Criteria:

* Positive serology for hepatitis B, hepatitis C, HIV, syphilis, HTLV-1
* Current or past medical disease that could interfere with the evaluation of the efficacy, as judged by the investigator
* Severe renal or hepatic impairment

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Cell biodistribution after intravenous infusion as assessed by SPECT/CT scan | 72 hours
Potential occurrence of any AE or SAE, related to the product, using patient open non-directive questionnaire, physical examination and laboratory measurements | 12 months

SECONDARY OUTCOMES:
Pain measured by the Visual Analogue Scale | 12 months
Well-being score using SF-36 questionnaire | 12 months
Occurrence of new vertebral fractures as assessed by X-ray | 12 months
Bone mineral density evolution as assessed by Dual-energy X-ray absorptiometry (DEXA) | 12 months
Measurement of bone formation and resorption markers | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Investigating site BE01, Anderlecht, Belgium